CLINICAL TRIAL: NCT03239431
Title: A 3 Year Longitudinal Study of the Level of Asthma Control and Treatment of Asthma Patients in Hong Kong
Brief Title: A Study to Determine the Clinical Characteristics, Comorbidities, Treatment Status and Exacerbations of Asthma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Honorary Clinical Tutor, Chinese University of Hong Kong
Other Study IDs: CREC 2017.336
Record Dates: First submitted 2017-07-27; First posted 2017-08-04 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: asthma; lung function; forced oscillometry technique; exacerbation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Genetic markers in blood sample that can help to predict exacerbation and level of control in patients with asthma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma group: Patients with asthma
  Interventions: Other: asthmatic exacerbation

INTERVENTIONS:
Other: asthmatic exacerbation — evaluate the risk factors, frequency and nature of asthma exacerbations

SUMMARY:
This is a prospective cohort study that aims to determine the current demographics, clinical characteristics, comorbidities, treatment status and exacerbations of asthma patients.

The primary objective of this study is to determine the current demographics, clinical characteristics, comorbidities, treatment status and exacerbations of asthma patients.

The secondary objectives include: (1) to review the current practices of symptom control assessment, (2) to determine the choice of pharmacological regimen, rate of guideline adherence and real-world clinical practice in managing asthma patients, (3) to evaluate the pattern of lung function parameters (spirometry and forced oscillometry technique [FOT]) in adult asthma patients, (4) to evaluate the effect of ageing on the trend of change in lung function parameters (spirometry and FOT) in adult asthma patients, (5) to identify biomarkers that help to categorize different asthma phenotypes and predict subsequent prognosis, (6) to determine the risk factors of uncontrolled asthma and asthma exacerbation, (7) to evaluate the impact of comorbidities on asthma control.

400 out-patient asthma patients are planned to be recruited and they will be followed up for 3 years.

DETAILED DESCRIPTION:
Asthma is a common respiratory disease worldwide and in Hong Kong. According to the estimation by the Center for Disease Control and Prevention in 2015, 7.6% adults in the United States have asthma. In Hong Kong, the prevalence of asthma was estimated to be 10.1% among 13 to 14 years old children and 5.8% in randomly selected Chinese elderly aged more than 70. With a rising trend of life expectancy in Hong Kong, the epidemiology of asthma in adult and elderly population may change over time. In addition, elderly patients with asthma may present with a different spectrum of clinical characteristics and pharmacological response.

Asthmatic exacerbation is one of the untoward complications and hospitalization for exacerbations requiring ICU care and mechanical ventilation are both predictors for near-fatal asthma. After the acute attack, its unfavourable impact continues and can lead to multiple sequelae. Exacerbation of asthma is associated with a more rapid decline in the post-bronchodilator forced expiratory volume in 1 second and worse quality of life. Without adjustment of medical treatment, they are prone to develop another episode of exacerbation within a short period of time. In addition, individuals with uncontrolled asthma had higher medical expenditures and decreased productivity, contributing to a greater economic burden when compared with individuals without asthma. In contrary, patients with controlled asthma had lower hospitalization rate, mortality rate and less lung function decline. Many risk factors for exacerbation had been identified including upper airway diseases, gastroesophageal reflux, poor inhaler technique, medication non-compliance. Many of these factors are potentially reversible. A model of better asthma care may be established by improving the understanding on these risk factors, leading to less exacerbation events.

Asthma is not simply an airway disease. Accumulating evidence showed its coexistence with other upper airway and systemic diseases, both atopic and non-atopic. These comorbidities independently or linked together to impose negative impact on patients' health status and quality of life. Knowing about the burden of asthma related comorbidities may help to guide clinician in managing these complications in a more effective way, and even prediction of subsequent prognosis.

Since the launching of GINA guideline in year 1993, its regular evidence-based update on pharmacological treatment had revolutionize the care of asthma patients. The use of asthma medications by both specialists and primary care physicians became more structured and the asthma control was improved. However, there is still a significant proportion of asthma patients experiencing recurrent exacerbation despite optimization of pharmacological treatment. Both the guideline adherence by physicians and drug compliance by patient are subjects of concern.

Previous evidence showed that the compliance rate of GINA guideline is far from satisfactory, which is a shared phenomenon among different common diseases even the presence of well-established international guideline. Patient's drug compliance also contributes to negative disease outcome, especially non-adherence to inhaled corticosteroid. Currently, a comprehensive view on the treatment status in and level of asthma control in Hong Kong is still lacking.

A large knowledge gap exists between the current demographics, comorbidities, treatment status, level of asthma control and exacerbations in Hong Kong. An updated study on these aspects is definitely warranted to enhance patient care and guide further research.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with confirmed diagnosis of asthma (defined as those with a consistent history and prior documented evidence of variable airflow obstruction, with evidence of an increase in FEV1 greater than 12% or 200 mL following bronchodilator or bronchial hyperresponsiveness on bronchial provocation testing, when stable (reference)
2. Age greater than 18 years old
3. Signed written informed consent to participate in the study

Exclusion Criteria:

1. Patients currently with acute exacerbation of asthma by GINA guideline (they can join the study after 6 weeks post recovery from the exacerbation)
2. Patients with respiratory diseases that can show similar symptoms to asthma such as bronchiectasis, tuberculosis-destroyed lung parenchyma, endobronchial TB, and lung cancer, or those who have history of these diseases based on physician's judgment
3. Patients with respiratory diseases that may confound the lung function parameters such as pleural diseases, interstitial lung diseases, and previous lung surgery, or those who have history of these diseases based on physician's judgment
4. Patients with neuromuscular diseases that may affect the seal off the mouthpiece during spirometry and forced oscillometry technique (FOT)
5. Patients with uncontrolled or active contagious respiratory infection diseases
6. Patients with smoking history more than 10 pack years
7. Significant comorbid illnesses that limit the life expectancy to less than 1 year
8. Patients who are mentally not fit or physically contraindicated for spirometry and FOT
9. Patients with psychiatric disease or cognitive impairment that may limit their ability of understanding or giving consent to the study
10. Patients currently randomized in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from the medical out-patient clinic by the physicians in the Prince of Wales Hospital. As the physicians will both attend general medical clinics and respiratory clinics, they will recruit patients from these clinics
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
The clinical characteristics of asthma patients | over 3 years
  The clinical characteristics of asthma patients
The treatment status of asthma patients | over 3 years
  The treatment status of asthma patients

SECONDARY OUTCOMES:
The 3 year morbidity of asthma patients | over 3 years
  The 3 year morbidity of asthma patients
The 3 year mortality of asthma patients | over 3 years
  The 3 year mortality of asthma patients
Genetic markers that predict exacerbation | over 3 years
  Genetic markers in blood sample that can help to predict exacerbation and level of control in patients with asthma

CONTACTS AND LOCATIONS:
Overall Officials: Ka Pang Chan, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: upon individual approach for metaanalysis or related study

REFERENCES:
- [Background] Wong GW, Leung TF, Ko FW. Changing prevalence of allergic diseases in the Asia-pacific region. Allergy Asthma Immunol Res. 2013 Sep;5(5):251-7. doi: 10.4168/aair.2013.5.5.251. Epub 2013 Mar 18. PMID 24003381
- [Background] Ko FW, Lai CK, Woo J, Ho SC, Ho CW, Goggins W, Hui DS. 12-year change in prevalence of respiratory symptoms in elderly Chinese living in Hong Kong. Respir Med. 2006 Sep;100(9):1598-607. doi: 10.1016/j.rmed.2005.12.007. Epub 2006 Jan 30. PMID 16446081
- [Background] Pasha MA, Sundquist B, Townley R. Asthma pathogenesis, diagnosis, and management in the elderly. Allergy Asthma Proc. 2017 May 1;38(3):184-191. doi: 10.2500/aap.2017.38.4048. PMID 28441988
- [Background] Serrano-Pariente J, Plaza V. Near-fatal asthma: a heterogeneous clinical entity. Curr Opin Allergy Clin Immunol. 2017 Feb;17(1):28-35. doi: 10.1097/ACI.0000000000000333. PMID 27870665
- [Background] Turner MO, Noertjojo K, Vedal S, Bai T, Crump S, Fitzgerald JM. Risk factors for near-fatal asthma. A case-control study in hospitalized patients with asthma. Am J Respir Crit Care Med. 1998 Jun;157(6 Pt 1):1804-9. doi: 10.1164/ajrccm.157.6.9708092. PMID 9620909
- [Background] Bai TR, Vonk JM, Postma DS, Boezen HM. Severe exacerbations predict excess lung function decline in asthma. Eur Respir J. 2007 Sep;30(3):452-6. doi: 10.1183/09031936.00165106. Epub 2007 May 30. PMID 17537763
- [Background] O'Byrne PM, Pedersen S, Lamm CJ, Tan WC, Busse WW; START Investigators Group. Severe exacerbations and decline in lung function in asthma. Am J Respir Crit Care Med. 2009 Jan 1;179(1):19-24. doi: 10.1164/rccm.200807-1126OC. Epub 2008 Oct 31. PMID 18990678
- [Background] Luskin AT, Chipps BE, Rasouliyan L, Miller DP, Haselkorn T, Dorenbaum A. Impact of asthma exacerbations and asthma triggers on asthma-related quality of life in patients with severe or difficult-to-treat asthma. J Allergy Clin Immunol Pract. 2014 Sep-Oct;2(5):544-52.e1-2. doi: 10.1016/j.jaip.2014.02.011. Epub 2014 Jul 3. PMID 25213047
- [Background] Miller MK, Lee JH, Miller DP, Wenzel SE; TENOR Study Group. Recent asthma exacerbations: a key predictor of future exacerbations. Respir Med. 2007 Mar;101(3):481-9. doi: 10.1016/j.rmed.2006.07.005. Epub 2006 Aug 17. PMID 16914299
- [Background] Sullivan PW, Slejko JF, Ghushchyan VH, Sucher B, Globe DR, Lin SL, Globe G. The relationship between asthma, asthma control and economic outcomes in the United States. J Asthma. 2014 Sep;51(7):769-78. doi: 10.3109/02770903.2014.906607. Epub 2014 Apr 7. PMID 24697738
- [Background] Moorman JE, Akinbami LJ, Bailey CM, Zahran HS, King ME, Johnson CA, Liu X. National surveillance of asthma: United States, 2001-2010. Vital Health Stat 3. 2012 Nov;(35):1-58. PMID 24252609
- [Background] ten Brinke A, Sterk PJ, Masclee AA, Spinhoven P, Schmidt JT, Zwinderman AH, Rabe KF, Bel EH. Risk factors of frequent exacerbations in difficult-to-treat asthma. Eur Respir J. 2005 Nov;26(5):812-8. doi: 10.1183/09031936.05.00037905. PMID 16264041
- [Background] Engelkes M, Janssens HM, de Jongste JC, Sturkenboom MC, Verhamme KM. Medication adherence and the risk of severe asthma exacerbations: a systematic review. Eur Respir J. 2015 Feb;45(2):396-407. doi: 10.1183/09031936.00075614. Epub 2014 Oct 16. PMID 25323234
- [Background] Tay TR, Radhakrishna N, Hore-Lacy F, Smith C, Hoy R, Dabscheck E, Hew M. Comorbidities in difficult asthma are independent risk factors for frequent exacerbations, poor control and diminished quality of life. Respirology. 2016 Nov;21(8):1384-1390. doi: 10.1111/resp.12838. Epub 2016 Jul 1. PMID 27363539
- [Background] Boulet LP. Influence of comorbid conditions on asthma. Eur Respir J. 2009 Apr;33(4):897-906. doi: 10.1183/09031936.00121308. PMID 19336592
- [Background] Robinson DS, Campbell DA, Durham SR, Pfeffer J, Barnes PJ, Chung KF; Asthma and Allergy Research Group of the National Heart and Lung Institute. Systematic assessment of difficult-to-treat asthma. Eur Respir J. 2003 Sep;22(3):478-83. doi: 10.1183/09031936.03.00017003. PMID 14516138
- [Background] Heaney LG, Conway E, Kelly C, Johnston BT, English C, Stevenson M, Gamble J. Predictors of therapy resistant asthma: outcome of a systematic evaluation protocol. Thorax. 2003 Jul;58(7):561-6. doi: 10.1136/thorax.58.7.561. PMID 12832665
- [Background] Bousquet J, Clark TJ, Hurd S, Khaltaev N, Lenfant C, O'byrne P, Sheffer A. GINA guidelines on asthma and beyond. Allergy. 2007 Feb;62(2):102-12. doi: 10.1111/j.1398-9995.2006.01305.x. PMID 17298416
- [Background] Dexheimer JW, Borycki EM, Chiu KW, Johnson KB, Aronsky D. A systematic review of the implementation and impact of asthma protocols. BMC Med Inform Decis Mak. 2014 Sep 9;14:82. doi: 10.1186/1472-6947-14-82. PMID 25204381
- [Background] Guarnaccia S, Lombardi A, Gaffurini A, Chiarini M, Domenighini S, D'Agata E, Schumacher RF, Spiazzi R, Notarangelo LD. Application and implementation of the GINA asthma guidelines by specialist and primary care physicians: a longitudinal follow-up study on 264 children. Prim Care Respir J. 2007 Dec;16(6):357-62. doi: 10.3132/pcrj.2007.00077. PMID 18038103
- [Background] Hekking PW, Wener RR, Amelink M, Zwinderman AH, Bouvy ML, Bel EH. The prevalence of severe refractory asthma. J Allergy Clin Immunol. 2015 Apr;135(4):896-902. doi: 10.1016/j.jaci.2014.08.042. Epub 2014 Oct 16. PMID 25441637
- [Background] Koga T, Oshita Y, Kamimura T, Koga H, Aizawa H. Characterisation of patients with frequent exacerbation of asthma. Respir Med. 2006 Feb;100(2):273-8. doi: 10.1016/j.rmed.2005.05.017. Epub 2005 Jul 5. PMID 15998585
- [Background] Scribano PV, Lerer T, Kennedy D, Cloutier MM. Provider adherence to a clinical practice guideline for acute asthma in a pediatric emergency department. Acad Emerg Med. 2001 Dec;8(12):1147-52. doi: 10.1111/j.1553-2712.2001.tb01131.x. PMID 11733292
- [Background] Shiffman RN, Freudigman Md, Brandt CA, Liaw Y, Navedo DD. A guideline implementation system using handheld computers for office management of asthma: effects on adherence and patient outcomes. Pediatrics. 2000 Apr;105(4 Pt 1):767-73. doi: 10.1542/peds.105.4.767. PMID 10742318
- [Background] Nestor A, Calhoun AC, Dickson M, Kalik CA. Cross-sectional analysis of the relationship between national guideline recommended asthma drug therapy and emergency/hospital use within a managed care population. Ann Allergy Asthma Immunol. 1998 Oct;81(4):327-30. doi: 10.1016/S1081-1206(10)63124-9. PMID 9809496
- [Background] Williams LK, Peterson EL, Wells K, Ahmedani BK, Kumar R, Burchard EG, Chowdhry VK, Favro D, Lanfear DE, Pladevall M. Quantifying the proportion of severe asthma exacerbations attributable to inhaled corticosteroid nonadherence. J Allergy Clin Immunol. 2011 Dec;128(6):1185-1191.e2. doi: 10.1016/j.jaci.2011.09.011. Epub 2011 Oct 21. PMID 22019090
- See also: CDC information on asthma. Assessed on 28 April 2017 — https://www.cdc.gov/asthma/most_recent_data.htm